CLINICAL TRIAL: NCT06836141
Title: Silent Brain Infarcts in Spontaneous Intracerebral Hemorrhage as a Prognostic Biomarker for Vascular Contributions to Cognitive Impairment and Dementia (VCID)
Brief Title: Biomarkers for Cognitive Decline in Intracerebral Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23022401; 1R01NS135614-01A1 (NIH)
Record Dates: First submitted 2025-01-15; First posted 2025-02-20 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Primary Intracerebral Hemorrhage
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — MRI during hospitalization and at 12 months post sICH
Diagnostic Test: Blood Draw — Will occur during hospitalization and at 3, 6 and 12 months post sICH
Diagnostic Test: Cognitive Test — Cognitive testing will occur during hospitalization and at 3, 6 and 12 months post sICH

SUMMARY:
The goal of this clinical trial is to see if silent brain infarcts (SBIs), or stroke-like symptoms detectable during brain imaging, are a possible contributor to cognitive decline for patients diagnosed with spontaneous intracerebral hemorrhage (sICH), or blood clot in the brain. The main questions it aims to answer are

* if SBIs in sICH are associated with a lower cognitive level and more rapid cognitive decline
* if SBIs in sICH are associated with certain findings on brain imaging
* if SBIs in sICH are associated with higher inflammation measured by certain blood tests

Participants will undergo

* cognitive testing during hospitalization, and at 3, 6 and 12 months after the sICH
* Magnetic Resonance Imaging (MRI) of the brain during hospitalization and 12 months after the sICH
* blood draws during hospitalization and at 3, 6 and 12 months after the sICH

DETAILED DESCRIPTION:
This proposal's objective is to establish SBIs (silent brain infarct) as an early, pathophysiologically plausible neuroimaging biomarker for VCID (vascular contributions to cognitive impairment and dementia) in sICH (spontaneous intracerebral hemorrhage) patients. To attain the overall objective, we will recruit a cohort of 118 sICH participants over 3 years and longitudinally measure cognitive function, WMH volumetric progression, and serum suPAR levels. Aim #1: To test the hypothesis that SBIs in sICH are associated with a lower cognitive level and more rapid cognitive decline. Approach: In sICH patients with and without SBIs, we will compare global cognition (primary analysis) and multiple cognitive domains (secondary analysis) at hospitalization, and at 3 months, 6 months, and 12 months after discharge using a comprehensive cognitive battery. Aim #2: To test the hypothesis that SBIs in sICH are associated with more rapid WMH (white matter hyperintensities) progression as measured by serial MRI (magnetic resonance imaging). Approach: In sICH patients with and without SBIs, we will compare the absolute volumetric change in WMH using a novel imaging analysis algorithm on serial 3-Tesla brain MRI at hospitalization and at 12 months after discharge. Aim #3: To test the hypothesis that SBIs in sICH are associated with higher chronic systemic inflammation as measured by serum suPAR. Approach: In sICH patients with and without SBIs, we will compare serum levels of suPAR at hospitalization, and at 3 months, 6 months, and 12 months after discharge.

This study will be a prospective longitudinal study of sICH patients comparing those with and without SBIs. All patients with primary sICH are admitted to Rush University Medical Center's (RUMC) Neurosciences Intensive Care Unit and managed by a multi-disciplinary team of neurologists and neurosurgeons according to a standardized protocol based on current guidelines. Primary sICH will be defined as either hypertensive or related to cerebral amyloid angiopathy as diagnosed using the Boston Criteria version 2.0. This differs from secondary sICH, defined as hemorrhage due to vascular malformation, coagulopathy, trauma, malignancy, or reversible vasculopathy. Before hospital discharge, participants will receive baseline cognitive testing, MRI brain, and suPAR (soluble urokinase-type plasminogen activator receptor) serology sampling. After discharge from the hospital, participants will follow up in RUMC's Comprehensive Stroke Clinic at 3 months as part of their routine stroke care per our center's protocol. At the 3-month visit, participants will receive cognitive testing and provide suPAR serology. Participants will complete an interim 6-month visit with cognitive testing and suPAR serology. At a 12-month research clinic visit, participants will repeat cognitive testing, brain MRI, and suPAR serology. All participant encounters will provide the opportunity to gather interim clinical data such as new medical diagnoses or repeat hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Primary Intracerebral Hemorrhage
* Age ≥ 18 and < 80 years

Exclusion Criteria:

* ICH score > 2
* Pre-existing dementia
* Prior history of stroke
* Neurosurgical evacuation of hematoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Rush University Medical Center with an intracerebral hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Global Cognition | From date of randomization and assessed throughout the during hospitalization for qualifying ICH event up to 12 months
  Assessed via the the Late Onset Alzheimer's Disease Family Study Cognitive Battery
Global Cognition | 3 months after hospitalization
  Assessed via the the Late Onset Alzheimer's Disease Family Study Cognitive Battery
Global Cognition | 6 months after hospitalization
  Assessed via the the Late Onset Alzheimer's Disease Family Study Cognitive Battery
Global Cognition | 12 months after hospitalization
  Assessed via the the Late Onset Alzheimer's Disease Family Study Cognitive Battery
Absolute volumetric change in White Matter Hyperintensity (WMH) | from MRI at hospitalization to MRI at 12 months
  Uses a novel imaging analysis algorithm on serial 3-Tesla brain MRI
Serum soluble urokinase-type plasminogen activator receptor (suPAR) levels | From date of consent and assessed during hospitalization for qualifying ICH event up to 12 months
  compare SuPAR levels between the silent brain infarct (SBI) positive and the SBI negative groups
Serum soluble urokinase-type plasminogen activator receptor (suPAR) levels | 3 months after hospital discharge
  compare SuPAR levels between the silent brain infarct (SBI) positive and the SBI negative
Serum soluble urokinase-type plasminogen activator receptor (suPAR) levels | 6 months after hospital discharge
  compare SuPAR levels between the silent brain infarct (SBI) positive and the SBI negative
Serum soluble urokinase-type plasminogen activator receptor (suPAR) levels | 12 months after hospital discharge
  compare SuPAR levels between the silent brain infarct (SBI) positive and the SBI negative

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Garg, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg SM, Ziai WC, Cordonnier C, Dowlatshahi D, Francis B, Goldstein JN, Hemphill JC 3rd, Johnson R, Keigher KM, Mack WJ, Mocco J, Newton EJ, Ruff IM, Sansing LH, Schulman S, Selim MH, Sheth KN, Sprigg N, Sunnerhagen KS; American Heart Association/American Stroke Association. 2022 Guideline for the Management of Patients With Spontaneous Intracerebral Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2022 Jul;53(7):e282-e361. doi: 10.1161/STR.0000000000000407. Epub 2022 May 17. No abstract available. PMID 35579034
- [Background] Hemorrhagic Stroke Academia Industry (HEADS) Roundtable Participants; Second HEADS Roundtable Participants. Recommendations for Clinical Trials in ICH: The Second Hemorrhagic Stroke Academia Industry Roundtable. Stroke. 2020 Apr;51(4):1333-1338. doi: 10.1161/STROKEAHA.119.027882. Epub 2020 Feb 10. No abstract available. PMID 32078490
- [Background] Hwang DY, Kim KS, Muehlschlegel S, Wartenberg KE, Rajajee V, Alexander SA, Busl KM, Creutzfeldt CJ, Fontaine GV, Hocker SE, Madzar D, Mahanes D, Mainali S, Sakowitz OW, Varelas PN, Weimar C, Westermaier T, Meixensberger J. Guidelines for Neuroprognostication in Critically Ill Adults with Intracerebral Hemorrhage. Neurocrit Care. 2024 Apr;40(2):395-414. doi: 10.1007/s12028-023-01854-7. Epub 2023 Nov 3. PMID 37923968
- [Background] Smith HW, Marshall CJ. Regulation of cell signalling by uPAR. Nat Rev Mol Cell Biol. 2010 Jan;11(1):23-36. doi: 10.1038/nrm2821. PMID 20027185
- [Background] Nikorowitsch J, Borchardt T, Appelbaum S, Ojeda F, Lackner KJ, Schnabel RB, Blankenberg S, Zeller T, Karakas M. Cardio-Renal Biomarker Soluble Urokinase-Type Plasminogen Activator Receptor Is Associated With Cardiovascular Death and Myocardial Infarction in Patients With Coronary Artery Disease Independent of Troponin, C-Reactive Protein, and Renal Function. J Am Heart Assoc. 2020 Apr 21;9(8):e015452. doi: 10.1161/JAHA.119.015452. Epub 2020 Apr 17. PMID 32299288
- [Background] Wilson RS, Yu L, Lamar M, Schneider JA, Boyle PA, Bennett DA. Education and cognitive reserve in old age. Neurology. 2019 Mar 5;92(10):e1041-e1050. doi: 10.1212/WNL.0000000000007036. Epub 2019 Feb 6. PMID 30728309
- [Background] Garg RK, Khan J, Dawe RJ, Conners J, John S, Prabhakaran S, Kocak M, Bhabad S, Simpson SL, Ouyang B, Jhaveri M, Bleck TP. The Influence of Diffusion Weighted Imaging Lesions on Outcomes in Patients with Acute Spontaneous Intracerebral Hemorrhage. Neurocrit Care. 2020 Oct;33(2):552-564. doi: 10.1007/s12028-020-00933-3. PMID 32072457
- [Background] Grosu S, Rospleszcz S, Hartmann F, Habes M, Bamberg F, Schlett CL, Galie F, Lorbeer R, Auweter S, Selder S, Buelow R, Heier M, Rathmann W, Mueller-Peltzer K, Ladwig KH, Grabe HJ, Peters A, Ertl-Wagner BB, Stoecklein S. Associated factors of white matter hyperintensity volume: a machine-learning approach. Sci Rep. 2021 Jan 27;11(1):2325. doi: 10.1038/s41598-021-81883-4. PMID 33504924
- [Background] Greenberg SM, O'Donnell HC, Schaefer PW, Kraft E. MRI detection of new hemorrhages: potential marker of progression in cerebral amyloid angiopathy. Neurology. 1999 Sep 22;53(5):1135-8. doi: 10.1212/wnl.53.5.1135. PMID 10496283
- [Background] Maclullich AM, Wardlaw JM, Ferguson KJ, Starr JM, Seckl JR, Deary IJ. Enlarged perivascular spaces are associated with cognitive function in healthy elderly men. J Neurol Neurosurg Psychiatry. 2004 Nov;75(11):1519-23. doi: 10.1136/jnnp.2003.030858. PMID 15489380
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Chew-Harris J, Appleby S, Richards AM, Troughton RW, Pemberton CJ. Analytical, biochemical and clearance considerations of soluble urokinase plasminogen activator receptor (suPAR) in healthy individuals. Clin Biochem. 2019 Jul;69:36-44. doi: 10.1016/j.clinbiochem.2019.05.010. Epub 2019 May 23. PMID 31129182
- [Background] Eugen-Olsen J, Ladelund S, Sorensen LT. Plasma suPAR is lowered by smoking cessation: a randomized controlled study. Eur J Clin Invest. 2016 Apr;46(4):305-11. doi: 10.1111/eci.12593. Epub 2016 Feb 19. PMID 26799247
- [Background] Haupt TH, Kallemose T, Ladelund S, Rasmussen LJ, Thorball CW, Andersen O, Pisinger C, Eugen-Olsen J. Risk factors associated with serum levels of the inflammatory biomarker soluble urokinase plasminogen activator receptor in a general population. Biomark Insights. 2014 Dec 16;9:91-100. doi: 10.4137/BMI.S19876. eCollection 2014. PMID 25574132
- [Background] Mehta A, Desai SR, Ko YA, Liu C, Dhindsa DS, Nayak A, Hooda A, Martini MA, Ejaz K, Sperling LS, Reiser J, Hayek SS, Quyyumi AA. Sex Differences in Circulating Soluble Urokinase-Type Plasminogen Activator Receptor (suPAR) Levels and Adverse Outcomes in Coronary Artery Disease. J Am Heart Assoc. 2020 Mar 3;9(5):e015457. doi: 10.1161/JAHA.119.015457. Epub 2020 Feb 22. PMID 32089048
- [Background] Chen X, Jin Y, Chen J, Chen X, Cao X, Yu L, Xu Y. Relationship between White Matter Hyperintensities and Hematoma Volume in Patients with Intracerebral Hematoma. Aging Dis. 2018 Dec 4;9(6):999-1009. doi: 10.14336/AD.2018.0108. eCollection 2018 Dec. PMID 30574413
- [Background] Dickie DA, Ritchie SJ, Cox SR, Sakka E, Royle NA, Aribisala BS, Valdes Hernandez Mdel C, Maniega SM, Pattie A, Corley J, Starr JM, Bastin ME, Deary IJ, Wardlaw JM. Vascular risk factors and progression of white matter hyperintensities in the Lothian Birth Cohort 1936. Neurobiol Aging. 2016 Jun;42:116-23. doi: 10.1016/j.neurobiolaging.2016.03.011. Epub 2016 Mar 21. PMID 27143428
- [Background] Zheng K, Wang Z, Chen X, Chen J, Fu Y, Chen Q. Analysis of Risk Factors for White Matter Hyperintensity in Older Adults without Stroke. Brain Sci. 2023 May 22;13(5):835. doi: 10.3390/brainsci13050835. PMID 37239307
- [Background] Scharf EL, Graff-Radford J, Przybelski SA, Lesnick TG, Mielke MM, Knopman DS, Preboske GM, Schwarz CG, Senjem ML, Gunter JL, Machulda M, Kantarci K, Petersen RC, Jack CR Jr, Vemuri P. Cardiometabolic Health and Longitudinal Progression of White Matter Hyperintensity: The Mayo Clinic Study of Aging. Stroke. 2019 Nov;50(11):3037-3044. doi: 10.1161/STROKEAHA.119.025822. Epub 2019 Sep 12. PMID 31510903
- [Background] Debette S, Seshadri S, Beiser A, Au R, Himali JJ, Palumbo C, Wolf PA, DeCarli C. Midlife vascular risk factor exposure accelerates structural brain aging and cognitive decline. Neurology. 2011 Aug 2;77(5):461-8. doi: 10.1212/WNL.0b013e318227b227. PMID 21810696
- [Background] van Dijk EJ, Prins ND, Vrooman HA, Hofman A, Koudstaal PJ, Breteler MM. Progression of cerebral small vessel disease in relation to risk factors and cognitive consequences: Rotterdam Scan study. Stroke. 2008 Oct;39(10):2712-9. doi: 10.1161/STROKEAHA.107.513176. Epub 2008 Jul 17. PMID 18635849
- [Background] Power MC, Deal JA, Sharrett AR, Jack CR Jr, Knopman D, Mosley TH, Gottesman RF. Smoking and white matter hyperintensity progression: the ARIC-MRI Study. Neurology. 2015 Feb 24;84(8):841-8. doi: 10.1212/WNL.0000000000001283. Epub 2015 Jan 28. PMID 25632094
- [Background] Posener S, Hmeydia G, Benzakoun J, Oppenheim C, Baron JC, Turc G. Remote Diffusion-Weighted Imaging Lesions and Intracerebral Hemorrhage: A Systematic Review and Meta-Analysis. Stroke. 2023 Apr;54(4):e133-e137. doi: 10.1161/STROKEAHA.122.040689. Epub 2023 Mar 3. PMID 36866676
- [Background] Bennett DA, De Jager PL, Leurgans SE, Schneider JA. Neuropathologic intermediate phenotypes enhance association to Alzheimer susceptibility alleles. Neurology. 2009 Apr 28;72(17):1495-503. doi: 10.1212/WNL.0b013e3181a2e87d. PMID 19398704
- [Background] Gong L, Gu Y, Yu Q, Wang H, Zhu X, Dong Q, Xu R, Zhao Y, Liu X. Prognostic Factors for Cognitive Recovery Beyond Early Poststroke Cognitive Impairment (PSCI): A Prospective Cohort Study of Spontaneous Intracerebral Hemorrhage. Front Neurol. 2020 Apr 28;11:278. doi: 10.3389/fneur.2020.00278. eCollection 2020. PMID 32411073
- [Background] Case NF, Charlton A, Zwiers A, Batool S, McCreary CR, Hogan DB, Ismail Z, Zerna C, Coutts SB, Frayne R, Goodyear B, Haffenden A, Smith EE. Cerebral Amyloid Angiopathy Is Associated With Executive Dysfunction and Mild Cognitive Impairment. Stroke. 2016 Aug;47(8):2010-6. doi: 10.1161/STROKEAHA.116.012999. Epub 2016 Jun 23. PMID 27338926
- [Background] Schmidt FA, Liotta EM, Prabhakaran S, Naidech AM, Maas MB. Assessment and comparison of the max-ICH score and ICH score by external validation. Neurology. 2018 Sep 4;91(10):e939-e946. doi: 10.1212/WNL.0000000000006117. Epub 2018 Aug 1. PMID 30068631
- [Background] Hemphill JC 3rd, Bonovich DC, Besmertis L, Manley GT, Johnston SC. The ICH score: a simple, reliable grading scale for intracerebral hemorrhage. Stroke. 2001 Apr;32(4):891-7. doi: 10.1161/01.str.32.4.891. PMID 11283388
- [Background] Pisani MA, Inouye SK, McNicoll L, Redlich CA. Screening for preexisting cognitive impairment in older intensive care unit patients: use of proxy assessment. J Am Geriatr Soc. 2003 May;51(5):689-93. doi: 10.1034/j.1600-0579.2003.00215.x. PMID 12752846
- [Background] Prabhakaran S, Gupta R, Ouyang B, John S, Temes RE, Mohammad Y, Lee VH, Bleck TP. Acute brain infarcts after spontaneous intracerebral hemorrhage: a diffusion-weighted imaging study. Stroke. 2010 Jan;41(1):89-94. doi: 10.1161/STROKEAHA.109.566257. Epub 2009 Nov 5. PMID 19892994
- [Background] Gupta A, Giambrone AE, Gialdini G, Finn C, Delgado D, Gutierrez J, Wright C, Beiser AS, Seshadri S, Pandya A, Kamel H. Silent Brain Infarction and Risk of Future Stroke: A Systematic Review and Meta-Analysis. Stroke. 2016 Mar;47(3):719-25. doi: 10.1161/STROKEAHA.115.011889. PMID 26888534
- [Background] Charidimou A, Boulouis G, Frosch MP, Baron JC, Pasi M, Albucher JF, Banerjee G, Barbato C, Bonneville F, Brandner S, Calviere L, Caparros F, Casolla B, Cordonnier C, Delisle MB, Deramecourt V, Dichgans M, Gokcal E, Herms J, Hernandez-Guillamon M, Jager HR, Jaunmuktane Z, Linn J, Martinez-Ramirez S, Martinez-Saez E, Mawrin C, Montaner J, Moulin S, Olivot JM, Piazza F, Puy L, Raposo N, Rodrigues MA, Roeber S, Romero JR, Samarasekera N, Schneider JA, Schreiber S, Schreiber F, Schwall C, Smith C, Szalardy L, Varlet P, Viguier A, Wardlaw JM, Warren A, Wollenweber FA, Zedde M, van Buchem MA, Gurol ME, Viswanathan A, Al-Shahi Salman R, Smith EE, Werring DJ, Greenberg SM. The Boston criteria version 2.0 for cerebral amyloid angiopathy: a multicentre, retrospective, MRI-neuropathology diagnostic accuracy study. Lancet Neurol. 2022 Aug;21(8):714-725. doi: 10.1016/S1474-4422(22)00208-3. PMID 35841910
- [Background] Jones WJ, Williams LS, Meschia JF. Validating the Questionnaire for Verifying Stroke-Free Status (QVSFS) by neurological history and examination. Stroke. 2001 Oct;32(10):2232-6. doi: 10.1161/hs1001.096191. PMID 11588306
- [Background] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170
- [Background] Wei C, El Hindi S, Li J, Fornoni A, Goes N, Sageshima J, Maiguel D, Karumanchi SA, Yap HK, Saleem M, Zhang Q, Nikolic B, Chaudhuri A, Daftarian P, Salido E, Torres A, Salifu M, Sarwal MM, Schaefer F, Morath C, Schwenger V, Zeier M, Gupta V, Roth D, Rastaldi MP, Burke G, Ruiz P, Reiser J. Circulating urokinase receptor as a cause of focal segmental glomerulosclerosis. Nat Med. 2011 Jul 31;17(8):952-60. doi: 10.1038/nm.2411. PMID 21804539
- [Background] Bifulco K, Longanesi-Cattani I, Gargiulo L, Maglio O, Cataldi M, De Rosa M, Stoppelli MP, Pavone V, Carriero MV. An urokinase receptor antagonist that inhibits cell migration by blocking the formyl peptide receptor. FEBS Lett. 2008 Apr 2;582(7):1141-6. doi: 10.1016/j.febslet.2008.03.001. Epub 2008 Mar 11. PMID 18339322
- [Background] Azam TU, Shadid HR, Blakely P, O'Hayer P, Berlin H, Pan M, Zhao P, Zhao L, Pennathur S, Pop-Busui R, Altintas I, Tingleff J, Stauning MA, Andersen O, Adami ME, Solomonidi N, Tsilika M, Tober-Lau P, Arnaoutoglou E, Keitel V, Tacke F, Chalkias A, Loosen SH, Giamarellos-Bourboulis EJ, Eugen-Olsen J, Reiser J, Hayek SS; International Study of Inflammation in COVID-19. Soluble Urokinase Receptor (SuPAR) in COVID-19-Related AKI. J Am Soc Nephrol. 2020 Nov;31(11):2725-2735. doi: 10.1681/ASN.2020060829. Epub 2020 Sep 22. PMID 32963090
- [Background] Botha S, Fourie CMT, Schutte R, Eugen-Olsen J, Pretorius R, Schutte AE. Soluble urokinase plasminogen activator receptor as a prognostic marker of all-cause and cardiovascular mortality in a black population. Int J Cardiol. 2015 Apr 1;184:631-636. doi: 10.1016/j.ijcard.2015.03.041. Epub 2015 Mar 4. PMID 25771228
- [Background] Persson M, Ostling G, Smith G, Hamrefors V, Melander O, Hedblad B, Engstrom G. Soluble urokinase plasminogen activator receptor: a risk factor for carotid plaque, stroke, and coronary artery disease. Stroke. 2014 Jan;45(1):18-23. doi: 10.1161/STROKEAHA.113.003305. Epub 2013 Nov 19. PMID 24253546
- [Background] Hayek SS, Leaf DE, Samman Tahhan A, Raad M, Sharma S, Waikar SS, Sever S, Camacho A, Wang X, Dande RR, Ibrahim NE, Baron RM, Altintas MM, Wei C, Sheikh-Hamad D, Pan JS, Holliday MW Jr, Januzzi JL, Weisbord SD, Quyyumi AA, Reiser J. Soluble Urokinase Receptor and Acute Kidney Injury. N Engl J Med. 2020 Jan 30;382(5):416-426. doi: 10.1056/NEJMoa1911481. PMID 31995687
- [Background] Hayek SS, Sever S, Ko YA, Trachtman H, Awad M, Wadhwani S, Altintas MM, Wei C, Hotton AL, French AL, Sperling LS, Lerakis S, Quyyumi AA, Reiser J. Soluble Urokinase Receptor and Chronic Kidney Disease. N Engl J Med. 2015 Nov 12;373(20):1916-25. doi: 10.1056/NEJMoa1506362. Epub 2015 Nov 5. PMID 26539835
- [Background] Timmermans K, Vaneker M, Scheffer GJ, Maassen P, Janssen S, Kox M, Pickkers P. Soluble urokinase-type plasminogen activator levels are related to plasma cytokine levels but have low predictive value for mortality in trauma patients. J Crit Care. 2015 Jun;30(3):476-80. doi: 10.1016/j.jcrc.2015.01.006. Epub 2015 Jan 9. PMID 25721031
- [Background] Lyngbaek S, Marott JL, Moller DV, Christiansen M, Iversen KK, Clemmensen PM, Eugen-Olsen J, Jeppesen JL, Hansen PR. Usefulness of soluble urokinase plasminogen activator receptor to predict repeat myocardial infarction and mortality in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous intervention. Am J Cardiol. 2012 Dec 15;110(12):1756-63. doi: 10.1016/j.amjcard.2012.08.008. Epub 2012 Sep 13. PMID 22981263
- [Background] Langkilde A, Jakobsen TL, Bandholm TQ, Eugen-Olsen J, Blauenfeldt T, Petersen J, Andersen O. Inflammation and post-operative recovery in patients undergoing total knee arthroplasty-secondary analysis of a randomized controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1265-1273. doi: 10.1016/j.joca.2017.03.008. Epub 2017 Mar 16. PMID 28323139
- [Background] Llinas P, Le Du MH, Gardsvoll H, Dano K, Ploug M, Gilquin B, Stura EA, Menez A. Crystal structure of the human urokinase plasminogen activator receptor bound to an antagonist peptide. EMBO J. 2005 May 4;24(9):1655-63. doi: 10.1038/sj.emboj.7600635. Epub 2005 Apr 7. PMID 15861141
- [Background] Biffi A, Bailey D, Anderson CD, Ayres AM, Gurol EM, Greenberg SM, Rosand J, Viswanathan A. Risk Factors Associated With Early vs Delayed Dementia After Intracerebral Hemorrhage. JAMA Neurol. 2016 Aug 1;73(8):969-76. doi: 10.1001/jamaneurol.2016.0955. PMID 27295605
- [Background] Moulin S, Labreuche J, Bombois S, Rossi C, Boulouis G, Henon H, Duhamel A, Leys D, Cordonnier C. Dementia risk after spontaneous intracerebral haemorrhage: a prospective cohort study. Lancet Neurol. 2016 Jul;15(8):820-829. doi: 10.1016/S1474-4422(16)00130-7. Epub 2016 Apr 28. PMID 27133238
- [Background] Schneider JA, Arvanitakis Z, Leurgans SE, Bennett DA. The neuropathology of probable Alzheimer disease and mild cognitive impairment. Ann Neurol. 2009 Aug;66(2):200-8. doi: 10.1002/ana.21706. PMID 19743450
- [Background] Schneider JA, Arvanitakis Z, Bang W, Bennett DA. Mixed brain pathologies account for most dementia cases in community-dwelling older persons. Neurology. 2007 Dec 11;69(24):2197-204. doi: 10.1212/01.wnl.0000271090.28148.24. Epub 2007 Jun 13. PMID 17568013
- [Background] Iadecola C, Duering M, Hachinski V, Joutel A, Pendlebury ST, Schneider JA, Dichgans M. Vascular Cognitive Impairment and Dementia: JACC Scientific Expert Panel. J Am Coll Cardiol. 2019 Jul 2;73(25):3326-3344. doi: 10.1016/j.jacc.2019.04.034. PMID 31248555
- [Background] Zlokovic BV, Gottesman RF, Bernstein KE, Seshadri S, McKee A, Snyder H, Greenberg SM, Yaffe K, Schaffer CB, Yuan C, Hughes TM, Daemen MJ, Williamson JD, Gonzalez HM, Schneider J, Wellington CL, Katusic ZS, Stoeckel L, Koenig JI, Corriveau RA, Fine L, Galis ZS, Reis J, Wright JD, Chen J. Vascular contributions to cognitive impairment and dementia (VCID): A report from the 2018 National Heart, Lung, and Blood Institute and National Institute of Neurological Disorders and Stroke Workshop. Alzheimers Dement. 2020 Dec;16(12):1714-1733. doi: 10.1002/alz.12157. Epub 2020 Oct 8. PMID 33030307
- [Background] Wilson RS, Leurgans SE, Foroud TM, Sweet RA, Graff-Radford N, Mayeux R, Bennett DA; National Institute on Aging Late-Onset Alzheimer's Disease Family Study Group. Telephone assessment of cognitive function in the late-onset Alzheimer's disease family study. Arch Neurol. 2010 Jul;67(7):855-61. doi: 10.1001/archneurol.2010.129. PMID 20625093

DOCUMENTS (1):
  • Informed Consent Form (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT06836141/ICF_000.pdf